CLINICAL TRIAL: NCT00280904
Title: A Registry for Comparing Catheter-Related Infection Rates Among Various Shunt Systems in the Treatment of Hydrocephalus
Status: Completed | Type: Observational
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Other Study IDs: CRI-IN04-001
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-02

CONDITIONS: Hydrocephalus
Keywords: Hydrocephalus; Shunt
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Shunt catheter — standard of care implantation of shunt (any brand). Subjects are followed for 90 days to obtain information about whether or not an infection occurred.

SUMMARY:
The purpose of this Registry is to compare shunt/catheter-related infection rates among various shunt systems when used according to hospital standard of care to treat hydrocephalus.

DETAILED DESCRIPTION:
Clinical trials show that the majority of infections in shunt systems originate from bacterial contamination introduced at the time of surgery and most appear by 3-4 weeks post-operatively. Protection must persist well beyond the surgical procedure to make certain that all contaminating bacteria are completely eradicated.

Depending upon the institution, shunt infection rates have been known to be as little as 1% to as much as 25%. However, two prospective trials that have been published from large databases, with a consistent definition of infection, have indicated an overall infection rate of approximately 10%

This prospective non-randomized, open-label Registry is designed to investigate and identify short-term shunt/catheter-related infection rates in ventriculoperitoneal shunt systems using various catheters during hospital standard of care treatment of Subjects with hydrocephalus. Prospective Subjects will include those receiving shunts for the first time (de novo) and those with previously implanted shunts for whom catheter or total system replacements are required.

This Registry will enroll 450 implanted Subjects of any age who meet all the inclusion criteria and none of the exclusion criteria and who provide signed Informed Consent to participate in this clinical Registry

Subjects will be followed for up to 90 days.

ELIGIBILITY:
Inclusion Criteria:

* The Subject requires a surgical procedure to implant (de novo) a ventriculoperitoneal shunt or to replace an already implanted shunt catheter for the treatment of hydrocephalus.
* The Subject (family member/legal representative) has completed the Informed Consent process prior to enrollment into this Registry.
* The Subject (family member/legal representative) is willing to comply with the Registry protocol timelines & requirements.

Exclusion Criteria:

* The Subject's planned shunt has distal drainage to the heart.
* The Subject has an active infection of the indwelling shunt system, cerebrospinal fluid or abdominal cavity.
* The Subject has ventriculitis, peritonitis or meningitis.
* The Subject has sepsis.
* The Subject has a history of poor wound healing.
* The Subject has symptoms pertaining to: a skin infection at or near the site of any incisions; an ear infection on either side; a respiratory tract infection; or a urinary tract infection that, in the Investigator's opinion is clinically significant and might compromise the outcome of this Registry.
* The Subject has had any form of bowel surgery 30 days prior to device implant or anticipates bowel surgery within 90 days following device implant
* The Subject has loculation(s) within the ventricular system.
* The Subject is otherwise determined by the Investigator to be medically unsuitable for participation in this Registry.
* The Subject is currently enrolled in another drug or device trial or has been previously entered in this trial.
* The Subject exhibits other difficulties, which would preclude follow-up for 90 days.
* The Subject is a prisoner.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects of any age, gender and ethnicity, with hydrocephalus
Sampling Method: Non-Probability Sample
Enrollment: 433 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Steinbok, MBBS, FRCSC, Study Chair — University of British Columbia
Locations (8):
- United States (2):
  - Children's memorial Hospital, Chicago, Illinois
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada
- China (2):
  - Prince of Wales Hospital, Beijing
  - Ua Shan Hospital, Shanghai
- Queen Mary Hospital, Hong Kong, Hong Kong
- All India Insitute of Medical Sciences, New Delhi, India
- National Neuroscience Institute, Singapore, Singapore

REFERENCES:
- [Result] Steinbok P, Milner R, Agrawal D, Farace E, Leung GK, Ng I, Tomita T, Wang E, Wang N, Wong GK, Zhou LF. A multicenter multinational registry for assessing ventriculoperitoneal shunt infections for hydrocephalus. Neurosurgery. 2010 Nov;67(5):1303-10. doi: 10.1227/NEU.0b013e3181f07e76. PMID 20871445

RESULTS

PARTICIPANT FLOW:
Groups:
- Ventriculoperitoneal Shunt Patients: Patients receiving a de novo standard or antibiotic (AI) catheter implant or catheter replacement of a prior ventriculoperitoneal shunt.
Period: Overall Study
Arm/Group | Ventriculoperitoneal Shunt Patients
Started | 433
Completed | 433
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ventriculoperitoneal Shunt Patients
Number analyzed (Participants) | 433
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 183
  Between 18 and 65 years | 193
  >=65 years | 57
Age Continuous [Mean (Standard Deviation); unit: years] | 31.3 (25.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194
  Male | 239

OUTCOME MEASURES:

1. Secondary Outcome: Non-infectious Antibiotic Impregnated (AI) and Standard Catheter Subjects With Shunt Failures
Time Frame: April 2008
Measure: Number; unit: participants
Groups:
- Ventriculoperitoneal Shunt Patients: Patients receiving a de novo antibiotic impregnated(AI)or standard catheter implant or catheter replacement of a prior ventriculoperitoneal shunt.
Arm/Group | Ventriculoperitoneal Shunt Patients
Number analyzed (Participants) | 433
participants | 40

2. Primary Outcome: Number of Subjects With Shunt Infections
Description: Number of shunt infections occurring in subjects implanted with antibiotic impregnated catheters and standard catheters.
Time Frame: Implantation to Explant
Measure: Number; unit: participants
Groups:
- Ventriculoperitoneal Shunt Patients: Patients receiving a de novo antibiotic impregnated (AI) or standard catheter implant or catheter replacement of a prior ventriculoperitoneal shunt.
Arm/Group | Ventriculoperitoneal Shunt Patients
Number analyzed (Participants) | 433
participants | 14

ADVERSE EVENTS:
Arm/Group | Ventriculoperitoneal Shunt Patients
Serious Adverse Events (participants affected / at risk) | 0/433
Other Adverse Events (participants affected / at risk) | 0/433

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less